CLINICAL TRIAL: NCT03408938
Title: The Value of Continuous Noninvasive Hemoglobin Monitoring Using Masimo Radical Pulse Co-oximeter in Intraoperative Blood Transfusion Practice During Obestatric Procedure
Brief Title: The Value of Continuous Noninvasive Hemoglobin Monitoring Using Masimo Radical -7 Pulse CO-Oximeter in Intraoperative Blood Transfusion Practice During Obstetric Procedures
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Ashraf Mohamed Abd Elmawgod (Unknown); Abdelhamid, Bassant Mohamed, M.D. (Individual); Hossam Eldin Mostafa Yahia (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia&I.C.U and Pain Clinic, Cairo University
Other Study IDs: N7-G1-2015/MD
Record Dates: First submitted 2017-12-29; First posted 2018-01-24 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Masimo Radical Pulse Co-oximeter in Intraoperative Blood Transfusion Practice During Obestatric Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Continuous Hb monitoring with Masimo Radical: Plethysmography Variability Index (PVI) is a measure of the dynamic changes in the perfusion index (PI) that occur during the respiratory cycle . PVI = ﴾PI Max - PI Min﴿ ÷ PI Maxx 100 %.
  PVI has the potential to provide useful information concerning changes in the balance between intrathoracic airway pressure and intravascular fluid volume. Trending of PVI may be useful in monitoring surgical patients, both intraoperatively and postoperatively, for appropriate hydration states. For example, a rising PVI may indicate developing hypovolemia and gives an alarm for the need of appropriate fluid and or blood products transfusion supported by the patient hemoglobin level
  Interventions: Device: of Masimo Radical-7¿ Pulse CO-Oximeter

INTERVENTIONS:
Device: of Masimo Radical-7¿ Pulse CO-Oximeter — The Masimo pulse oximetry model:
  The pulse oximetry model which Masimo developed accounts for saturation values contributed by the true arterial signal, and by one or more motion or noise signals. lt is assumed that under conditions of motion, the detected IR and RD signals comprise both the true arterial saturation signal and a venous (or non-arterial) motion noise signal. Masimo uses a highly sophisticated adaptive filter with, Discrete saturation transform (DST) four other parallel engines, to leverage each algorithm's unique strengths to ensure accurate readings through all patient conditions. Masimo SET's most powerful algorithm is Signal extraction technology (SET). All algorithms depend upon assumptions. The more assumptions, the weaker the algorithm. DST makes only one assumption -that arterial blood has a higher oxygenation than venous - making it the most powerful pulse oximetry algorithm
  Other Names: Puls Oximeter

SUMMARY:
The principle aim of this study is to detect the accurracy of Masimo Radical-7¿ Pulse CO-Oximeter in relation to laboratory hemoglobin and estimated blood loss in intraoperative blood transfusion practice during obstetric procedures with high risk of bleeding.

DETAILED DESCRIPTION:
Photoplethysmography of peripheral perfusion can be displayed by pulse oximeters. While the pulse oximeterplethysmogram represents a volume change and the arterial line blood pressure tracing represents a pressure change, it has been demonstrated that cyclical shifts in the plethysmogram reflect similar cyclic changes in the blood pressure tracing and that these changes reflect changes in the intravascular volume status of patients.Plethysmography Variability Index (PVI) is a measure of the dynamic changes in the perfusion index (PI) that occur during the respiratory cycle . PVI = ﴾PI Max - PI Min﴿ ÷ PI Maxx 100 %.

PVI has the potential to provide useful information concerning changes in the balance between intrathoracic airway pressure and intravascular fluid volume. Trending of PVI may be useful in monitoring surgical patients, both intraoperatively and postoperatively, for appropriate hydration states. For example, a rising PVI may indicate developing hypovolemia and gives an alarm for the need of appropriate fluid and or blood products transfusion supported by the patient hemoglobin level.

Continuous Hb monitoring may allow a more rapid detection of clinically significant blood loss, and has the potential to significantly improve perioperative transfusion practices, may enable a more rapid assessment of a patient's condition and more appropriate blood management and even perhaps reduce needless transfusions.

ELIGIBILITY:
Inclusion Criteria:

1. All adult high risk patients (ASA 1-2)
2. Age group (16-44 years old)
3. Obtetric surgery with high risk of bleeding in early and late pregnancy e.g Disturbed ectopic pregnancy ,Vesicular mole , Abortion , Placenta accrete , Rupture uterus and placenta previa

Exclusion Criteria:

1. Significant liver disease defined as (serum alanine aminotransferase and serum aspartate aminotransferase >2.5 times normal).
2. Significant renal disease defined as (serum creatinine >1.5 mg/dl or creatinine clearance <40 ml/min).
3. Significant coagulopathy defined as (INR >1.5).
4. Use of antiplatlets or anticoagulants.
5. Anemic patients with Hb% less than 8 gm/dl

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Basic subject demographics summary of age, weight, height, patient position, basal lab Hb, and start time of ADC. Basic summary of number of patients, estimated blood loss, transfusions, fluids given, mean arterial blood pressure, central venous pressure, fomites number and urine output.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Transfusion improvement | 24 hours
  Improvement of transfusion practice by detecting the amount of transfused units of RBCs during rapid blood loss

SECONDARY OUTCOMES:
Agreement between SpHb and laboratory Hb values | 24 hours
  The frequency of laboratory Hb testing and agreement between SpHb and laboratory Hb values

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Abdelmawgood, M.D, Study Chair — Professor of Anesthesia&I.C.U and Pain Clinic; Hossam El Din Mostafa, M.S, Study Director — Assistant Lecturer of Anesthesia&I.C.U and Pain Clinic
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Via scholar Gate